CLINICAL TRIAL: NCT06034795
Title: Evaluation of Bone Metabolism in Children and Adolescents With Familial Mediterranean Fever and Correlation With Genotype
Brief Title: Evaluation of Bone Metabolism in Children and Adolescents With Familial Mediterranean Fever
Acronym: FMF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Papageorgiou General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: q3e689cu
Record Dates: First submitted 2023-06-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Familial Mediterranean Fever
Keywords: Familial Mediterranean Fever; Bone mineral density; Low vitamin D; DEXA
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood samples will be tested for MEFV.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: 32 patients with Familial mediterranenan fever will participate. In these patients we will check bone mineral density using the dexa method.
  Blood tests will also be taken to assess calcium metabolism. All patients will be treated with colchicine.
- Control group: Healthy children will be used as control group. MEFV gene will be checked to exclude diagnosis of FMF. In these patients we will check bone mineral density using the dexa method. Blood tests will also be taken to assess calcium metabolism. The results from the two groups will be compared.

SUMMARY:
Familial Mediterranean Fever is a chronic auto-inflammatory disease. In the context of chronic inflammation, it seems that, among others, it also affects bone density in children. Bone loss may be due to subclinical inflammation that persists even during periods of remission. In addition, inflammatory cytokines also play an important role (mainly during episodes) resulting in an increase in bone degradation and ultimately a reduction in bone mass. Cytokines mainly associated with bone degradation and osteoclast activity are: IL-1R, IL-2, IL-6, IL-8, TNFa.

The purpose of this study is to determine the effect of FMF on bone density and to compare the results with a healthy population. In addition, the difference between the children with FMF will be studied according to the mutation they carry.

DETAILED DESCRIPTION:
For the above purpose, 62 children will participate, 31 healthy and 31 with FMF(confirmed mutation/s in the MEFV (Marenostrin Encoding Fever Gene) ).

They will be separated based on gender (boys, girls) and age: 2 age groups: a) 6-12 years, b) 12 - 20 years, separation into pre-adolescent children and adolescents (according to Tanner) and Body Mass Index ( BMI) (3rd-90th ED). Of the 31 children with FMF, all will be treated with colchicine and the study will not take place during periods of disease attack.

An attack free period is defined as a period of at least 3 weeks without clinical symptoms (fever, abdominal pain, arthritis) and without acute phase indicators (increased CRP, TKE, WBC).

The healthy population will exclude children with a history of disease related to a bone disorder. In addition, the existence of other factors that could affect bone density will be investigated in all 62 children. For this reason, there will be a check of calcium metabolism, vitamin D, kidney function, hormonal check, thyroid function check. Biomarkers of the RANK/RANKL/OPG axis that have a major role in osteoblast/osteoclast activity will be tested. Children's physical activity will be also assessed.

Bone density measurement will be done with a Hologic DISCOVERY QDR DXA (Dual Energy X-ray Absorptiometry) machine, the "gold standard" for spine and hip bone disorder screening worldwide. The program to be implemented will be adapted to childhood.

Then the following will be assessed: Body Mineral Density (BMD), Body Mineral Content (BMC) and z-score for the vertebrae of the OMSS (O1-O4) and Total Body less Head (TBLH).

ELIGIBILITY:
Inclusion Criteria:

* For patients:

  * Age > 6 years
  * BMI 3rd - 90th percentile
  * Meet the Tel Hashomer criteria (Avi Linhnen 1997)
  * Confirmed diagnosis by finding mutation(s) in the MEFV gene
  * Taking medication (colchicine) for at least 3 months
  * Normal physical activity during the last month, according to the questionnaire that will be distributed
  * Free individual history for bone diseases
  * Normal thyroid function
* For the control group:

  * Age > 6 years
  * BMI 3rd - 90th percentile
  * Free individual history for bone diseases
  * Normal physical activity according to the questionnaire
  * Normal thyroid function

Exclusion Criteria:

* For patients:

  * Age < 6 years
  * BMI < 3rd or > 90th percentile
  * Period of attack period of the disease
  * Those who have not started treatment with colchicine
  * Those who do not adapt well to taking colchicine
  * Decreased physical activity during the last month according to the questionnaire
  * Finding from the history of bone diseases that could affect the results
  * Taking vitamins that could affect the results
  * Existence of a factor that does not allow the performance of Dexa (when for example the safe and appropriate placement of the child cannot be ensured)
  * History of previous surgery which forced the patient to be bedridden for a significant period of time. Possible unreliable result of bone mineral density measurement due to reduced physical activity.
* For the control group:

  * Age < 6 years
  * BMI < 3rd or > 90th percentile
  * Taking vitamins that could affect the results
  * Decreased physical activity during the last month according to the questionnaire
  * History of previous surgery in the last year

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Two groups will be used: patients and control group. The results from blood examination and DEXA will be compared in order to check differences in bone mineral density betwwen the two groups.
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2022-01-08 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Effect of chronic inflammation of FMF on bone metabolism | The evaluation of bone mineral density will take place for children with FMF at attack free periods and for control group at periods that they are completely healthy. The maximun duration of the above control will be 24 hours.
  This study will include 62 children, 31 healthy and 31 with FMF.
  All children will undergo:
  1. Blood examination that will include check of calcium metabolism, Vitamin D levels, kidney function, hormonal control, thyroid function control. Biomarkers of the RANK/RANKL/OPG, which have a major role in osteoblast/osteoclast activity, will be tested.
  The subjects will be devided according to gender and age: 2 age groups: a) 6-12 years, b) 12 - 20 years.
  All the parameters will be compared to check if there is statistically significant difference between healthy children and children with FMF.
Effect of chronic inflammation of FMF on bone density | The evaluation of bone mineral density will take place for children with FMF at attack free periods and for control group at periods that they are completely healthy. The maximun duration of the above control will be 24 hours.
  All children will undergo:
  2. Bone density measurment by Dual Energy X-ray Absorptiometry (the most reliable method for imaging bone density and with the minimum radiation). We will check z-score of Lumbar spine and z-score of Total Body Less Head.
Effect of obesity on chronic inflammation of FMF | The evaluation of bone mineral density will take place for children with FMF at attack free periods and for control group at periods that they are completely healthy. The maximun duration of the above control will be 24 hours.
  We will measure Body Mass Index (BMI) in all subjects. We will measure weight in kilograms (kg) and height in meters (m) to arrive at one reported value of BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fotoulaki, Professor, Study Chair — Papageorgiou General Hospital; Effimia Papadopoulou, Professor, Study Director — Papageorgiou General Hospital; Christina Chaintari, Pediatrician, Principal Investigator — Papageorgiou General Hospital; Assimina Galli, Professor, Study Chair — AHEPA General Hospital
Locations (1):
- Papageorgiou General Hospital, Thessaloniki, Municipality of Pavlou Mela, Greece